CLINICAL TRIAL: NCT00839319
Title: Manipulation of the Intratesticular Hormonal Milieu With Exogenous Testosterone (Short Title (HOP-3)
Brief Title: HOP-3 Manipulation of the Intratesticular Hormonal Milieu With Exogenous Testosterone
Acronym: HOP-3
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, John Amory, Professor, Department of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27158-D; U54HD012629 (NIH)
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Results first posted 2010-11-16 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Healthy Males
Keywords: hCG; testosterone; Acyline; Intratesticular hormone
MeSH Terms: interventions — acyline; Chorionic Gonadotropin; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Acyline plus Placebo (Experimental): Acyline 300 ug/kg subcutaneous (SQ) injections on Day 1 plus subcutaneous placebo hCG injection (inj) every other day (5 doses) for 10 days
  Interventions: Drug: Acyline; Other: placebo hCG (no active ingredient)
- Acyline plus 15 IU hCG (Experimental): Acyline 300 ug/kg (SQ) inj(s) on Day 1 plus subcutaneous 15 IU hCG injection (inj) every other day (5 doses) for 10 days
  Interventions: Drug: Acyline; Drug: hCG (human chorionic gonadotropin)
- Acyline plus 60 IU hCG (Experimental): Acyline 300 ug/kg subcutaneous (SQ) injections on Day 1 plus subcutaneous 60 IU hCG injection (inj) every other day (5 doses) for 10 days
  Interventions: Drug: Acyline; Drug: hCG (human chorionic gonadotropin)
- Acyline plus 125 IU hCG (Experimental): Acyline 300 ug/kg subcutaneous (SQ) injections on Day 1 plus subcutaneous 125 IU hCG injection (inj) every other day (5 doses) for 10 days
  Interventions: Drug: Acyline; Drug: hCG (human chorionic gonadotropin)
- Acyline plus Testosterone gel (Experimental): Acyline 300 ug/kg subcutaneous (SQ) injections on Day 1 plus Testosterone gel 75 mg/day daily for 10 days
  Interventions: Drug: Acyline; Drug: Testosterone gel

INTERVENTIONS:
Drug: Acyline — 300 ug/kg subcutaneous injections on Day 1.
  Other Names: Acyline GhRH antagonist
Other: placebo hCG (no active ingredient) — placebo hCG
  Other Names: placebo drug
  Arms: Acyline plus Placebo
Drug: hCG (human chorionic gonadotropin) — 15 IU subcutaneous injection every other day for 10 days (5 doses)
  Other Names: Pregnyl
  Arms: Acyline plus 15 IU hCG
Drug: hCG (human chorionic gonadotropin) — 60 IU subcutaneous injection
  Other Names: Pregnyl
  Arms: Acyline plus 60 IU hCG
Drug: hCG (human chorionic gonadotropin) — 125 IU subcutaneous injection
  Other Names: Pregnyl
  Arms: Acyline plus 125 IU hCG
Drug: Testosterone gel — 75 mg testosterone gel applied transdermally for 10 days
  Other Names: Testim
  Arms: Acyline plus Testosterone gel

SUMMARY:
The purpose of this investigational study is to determine how much male hormone, testosterone, is necessary to maintain sperm production in the testis. This knowledge will be used to help in the development of a safe male hormonal contraception.

DETAILED DESCRIPTION:
Three study drugs will be used in this study: Testim (testosterone gel), Human Chorionic Gonadotropin (hCG) and acyline. Testosterone is a naturally occurring hormone in men. When given to normal men, testosterone gel will temporarily lower the amount of testosterone in the testes and lower sperm counts. hCG is a female hormone produced during pregnancy that is similar to and has the same actions as a male hormone, luteinizing hormone (LH). Like LH, hCG stimulates the testis to produce testosterone and sperm, and is used in the treatment of men who are deficient in LH. When hCG is given together with testosterone to normal men, the amount of testosterone in the testes will change, dependent on the amount of hCG received. Some participants will receive placebo hCG injections (no active medication).

Acyline suppresses LH (luteinizing hormone) and FSH (follicle stimulating hormone), which are hormones made by the pituitary gland in the brain, thus blocking the signal from the brain that causes the testes to make testosterone. Therefore, acyline blocks testosterone production. Men may experience some side effects from the low levels of testosterone caused by acyline.

Acyline is an experimental drug. Testosterone gel and hCG are approved for use in men with low testosterone levels. The U.S. Food and Drug Administration (FDA) allows testosterone gel, hCG and acyline to be given in combination for research to a small number of volunteers. Over 125 men have received acyline. Both Acyline and hCG will be given by injection. Acyline injections are formulated by subjects weight and may be given in multiple injections.

Participation will last approximately 2 months. The study involves a minimum of 9 visits in Seattle, WA. Clinic visits at Screening, Day 1 and Day 10 will take about 1-1.5 hours each. On Day 1 & 10 a fine needle aspiration of one testis will be performed. The Day 7, Day 17, and Day 40 visits will take approximately 30 minutes. The other visits will take about 15 minutes each time. Over the course of the study, which includes 5 separate blood draws, approximately 12 ounces (one and a half cups) of blood will be drawn. Some of the study drugs will be given by injection. One drug is a topical gel.

This is NOT a trial of a male contraceptive, and the study medications will not prevent pregnancy. Subjects must use an acceptable form of birth control.

ELIGIBILITY:
Inclusion Criteria:

* Males age 18-50
* Normal serum testosterone, LH and FSH
* PSA < 4.0
* Agrees not to donate blood or participate in another research study during the study
* Informed consent
* In general good health based on normal screening evaluation (consisting of a medical history, physical exam, normal sperm count, normal serum chemistry and hematology)
* Must be willing to use a reliable form of contraception during the study

Exclusion Criteria:

* Oligospermia (sperm count < 15 million/mL after 48 hours of abstinence) and/or abnormal motility or morphology.
* Participation in a long-term male contraceptive study within the past three months
* History of testosterone or anabolic steroid abuse in the past
* Poor general health with significantly abnormal blood results
* History of or current testicular disease
* History of a bleeding disorder or need for anticoagulation
* History of sleep apnea and/or major psychiatric problems
* BMI > 32
* Subjects with a skin condition that might interfere or be exacerbated by testosterone gel use
* Subject's with alcohol or drug use

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2009-03; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Bremner, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Contraceptive efficacy of testosterone-induced azoospermia in normal men. World Health Organization Task Force on methods for the regulation of male fertility. Lancet. 1990 Oct 20;336(8721):955-9. PMID 1977002
- [Background] Wu FC, Farley TM, Peregoudov A, Waites GM. Effects of testosterone enanthate in normal men: experience from a multicenter contraceptive efficacy study. World Health Organization Task Force on Methods for the Regulation of Male Fertility. Fertil Steril. 1996 Mar;65(3):626-36. PMID 8774299
- [Background] Anawalt BD, Bebb RA, Bremner WJ, Matsumoto AM. A lower dosage levonorgestrel and testosterone combination effectively suppresses spermatogenesis and circulating gonadotropin levels with fewer metabolic effects than higher dosage combinations. J Androl. 1999 May-Jun;20(3):407-14. PMID 10386821
- [Background] Zirkin BR, Santulli R, Awoniyi CA, Ewing LL. Maintenance of advanced spermatogenic cells in the adult rat testis: quantitative relationship to testosterone concentration within the testis. Endocrinology. 1989 Jun;124(6):3043-9. doi: 10.1210/endo-124-6-3043. PMID 2498065
- [Background] Coviello AD, Matsumoto AM, Bremner WJ, Herbst KL, Amory JK, Anawalt BD, Sutton PR, Wright WW, Brown TR, Yan X, Zirkin BR, Jarow JP. Low-dose human chorionic gonadotropin maintains intratesticular testosterone in normal men with testosterone-induced gonadotropin suppression. J Clin Endocrinol Metab. 2005 May;90(5):2595-602. doi: 10.1210/jc.2004-0802. Epub 2005 Feb 15. PMID 15713727
- [Background] Coviello AD, Bremner WJ, Matsumoto AM, Herbst KL, Amory JK, Anawalt BD, Yan X, Brown TR, Wright WW, Zirkin BR, Jarow JP. Intratesticular testosterone concentrations comparable with serum levels are not sufficient to maintain normal sperm production in men receiving a hormonal contraceptive regimen. J Androl. 2004 Nov-Dec;25(6):931-8. doi: 10.1002/j.1939-4640.2004.tb03164.x. PMID 15477366
- [Background] Awoniyi CA, Sprando RL, Santulli R, Chandrashekar V, Ewing LL, Zirkin BR. Restoration of spermatogenesis by exogenously administered testosterone in rats made azoospermic by hypophysectomy or withdrawal of luteinizing hormone alone. Endocrinology. 1990 Jul;127(1):177-84. doi: 10.1210/endo-127-1-177. PMID 2113863
- [Background] Chen H, Chandrashekar V, Zirkin BR. Can spermatogenesis be maintained quantitatively in intact adult rats with exogenously administered dihydrotestosterone? J Androl. 1994 Mar-Apr;15(2):132-8. PMID 8056636
- [Background] Meriggiola MC, Costantino A, Bremner WJ, Morselli-Labate AM. Higher testosterone dose impairs sperm suppression induced by a combined androgen-progestin regimen. J Androl. 2002 Sep-Oct;23(5):684-90. PMID 12185103
- [Result] Roth MY, Page ST, Lin K, Anawalt BD, Matsumoto AM, Snyder CN, Marck BT, Bremner WJ, Amory JK. Dose-dependent increase in intratesticular testosterone by very low-dose human chorionic gonadotropin in normal men with experimental gonadotropin deficiency. J Clin Endocrinol Metab. 2010 Aug;95(8):3806-13. doi: 10.1210/jc.2010-0360. Epub 2010 May 19. PMID 20484472
- [Result] Roth MY, Lin K, Bay K, Amory JK, Anawalt BD, Matsumoto AM, Marck BT, Bremner WJ, Page ST. Serum insulin-like factor 3 is highly correlated with intratesticular testosterone in normal men with acute, experimental gonadotropin deficiency stimulated with low-dose human chorionic gonadotropin: a randomized, controlled trial. Fertil Steril. 2013 Jan;99(1):132-139. doi: 10.1016/j.fertnstert.2012.09.009. Epub 2012 Oct 3. PMID 23040523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited using rosters from prior research studies and newspaper and online advertisements.
Pre-assignment Details: 2 of 61 men decided not to enroll. 19 failed inclusion criteria, 1 withdrew consent before study procedures, 1 dropped out after Day 1, and 1 was withdrawn by the investigator for syncopal reaction. 6 did not suppress serum luteinizing hormone(affecting intratesticular testosterone)and were excluded from analysis. 31 completed the study.
Groups:
- Acyline Plus Placebo: Acyline (ACY) 300 ug/kg subcutaneous (SQ) injections on Day 1 plus SQ placebo hCG every other day(q.o.d) (5 doses) for 10 days
- Acyline Plus 15 IU hCG: ACY 300 ug/kg SQ on Day 1 plus SQ 15 IU hCG q.o.d (5 doses) for 10 days
- Acyline Plus 60 IU hCG: ACY 300 ug/kg SQ Day 1 + 60 IU hCG SQ q.o.d (5 doses) for 10 days
- Acyline Plus 125 IU hCG: ACY 300 ug/kg SQ Day 1 + 125 IU hCG SQ q.o.d (5 doses) for 10 days
- Acyline Plus Testosterone Gel: ACY 300 ug/kg SQ on Day 1 + Testosterone gel 75 mg/day daily for 10 days
Period: Overall Study
Arm/Group | Acyline Plus Placebo | Acyline Plus 15 IU hCG | Acyline Plus 60 IU hCG | Acyline Plus 125 IU hCG | Acyline Plus Testosterone Gel
Started | 8 | 8 | 8 | 8 | 8
Completed | 6 (1 withdrew consent prior to procedures; 1 excluded from analysis (low serum LH)) | 7 (1 excluded from analysis (low serum LH)) | 5 (1 dropped out after Day 1 visit, 2 excluded from analysis (low serum LH)) | 5 (1 withdrawn by investigator for syncopal reaction , 2 excluded from analysis (low serum LH)) | 8
Not Completed | 2 | 1 | 3 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acyline Plus Placebo | Acyline Plus 15 IU hCG | Acyline Plus 60 IU hCG | Acyline Plus 125 IU hCG | Acyline Plus Testosterone Gel | Total
Number analyzed (Participants) | 6 | 7 | 5 | 5 | 8 | 31
Age, Customized [Median (Inter-Quartile Range); unit: years] | 21 [20 to 26] | 25 [20 to 29] | 22 [20 to 24] | 22 [21 to 26] | 22 [20 to 24] | 22 [20 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 7 | 5 | 5 | 8 | 31
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 24.8 [23.6 to 26.3] | 24.1 [23.2 to 26.7] | 24.9 [21.2 to 26.3] | 25.8 [22.9 to 26] | 23.7 [21.1 to 25.4] | 24.1 [22.9 to 26.3]
Serum Luteinizing Hormone (LH) [Median (Inter-Quartile Range); unit: IU/L] | 3.5 [3.1 to 4.8] | 3.0 [2.6 to 4.9] | 3.4 [3.4 to 4.9] | 2.9 [2.3 to 3.7] | 3.8 [2.6 to 4.6] | 3.4 [2.6 to 4.9]
Serum Follicle Simulating Hormone (FSH) [Median (Inter-Quartile Range); unit: IU/L] | 2.7 [1.2 to 3.4] | 2.4 [2 to 2.8] | 2.6 [2.2 to 3.2] | 2.2 [1.9 to 2.5] | 1.9 [1.3 to 2.8] | 2.4 [1.5 to 3.0]
Serum Testosterone (T) [Median (Inter-Quartile Range); unit: nmol/L] | 13.0 [11.3 to 16.9] | 15.0 [11.4 to 20.9] | 14.2 [12.7 to 14.9] | 16.8 [14.4 to 18.6] | 15.0 [13.7 to 18.3] | 14.6 [12 to 17.3]
Serum Dihydrotestosterone (DHT) [Median (Inter-Quartile Range); unit: nmol/L] | 1.0 [0.7 to 1.5] | 1.3 [0.9 to 1.7] | 1.2 [1 to 1.3] | 0.9 [0.7 to 1.5] | 1.1 [1.1 to 1.2] | 1.1 [0.9 to 1.4]
Serum Estradiol [Median (Inter-Quartile Range); unit: pmol/L] | 89 [47 to 150] | 65 [34 to 125] | 62 [48 to 78] | 77 [44 to 95] | 86 [54 to 95] | 77 [46 to 104]
Serum 17-Hydroxyprogesterone [Median (Inter-Quartile Range); unit: nmol/L] | 4.7 [3.8 to 7.8] | 4.9 [4.2 to 6.5] | 5.9 [5.1 to 7.6] | 4.3 [4 to 4.5] | 4.6 [3.7 to 5.4] | 4.9 [3.9 to 6.5]
Intratesticular Testosterone (ITT-T) [Median (Inter-Quartile Range); unit: nmol/L] | 3467 [2508 to 3839] | 2425 [1700 to 3380] | 1821 [1753 to 2412] | 3502 [2305 to 3959] | 2933 [1527 to 3390] | 2508 [1753 to 3502]
Intratesticular Dihydrotestosterone (ITT-DHT) [Median (Inter-Quartile Range); unit: nmol/L] | 18.0 [11.9 to 24.5] | 5.0 [4.5 to 11] | 7.6 [7.1 to 21.3] | 18.8 [11.1 to 22.2] | 12.9 [7.9 to 15.5] | 11.9 [7.3 to 21.3]

OUTCOME MEASURES:

1. Primary Outcome: Serum Testosterone (T)
Time Frame: 10 days
Population: Analysis per protocol. Due to nonnormality, the data were expressed as medians and 25th and 75 percentiles. Analysis of both baseline and end of treatment hormone concentrations performed on 31 subjects who completed all study procedures and who suppressed serum LH below the lower limit of normal at end of treatment.
Measure: Median (Inter-Quartile Range); unit: nmol/liter
Arm/Group | Acyline Plus Placebo | Acyline Plus 15 IU hCG | Acyline Plus 60 IU hCG | Acyline Plus 125 IU hCG | Acyline Plus Testosterone Gel
Number analyzed (Participants) | 6 | 7 | 5 | 5 | 8
nmol/liter | 0.43 [0.35 to 0.76] | 1.5 [0.79 to 4.9] | 3.7 [1 to 8.5] | 8.4 [4.9 to 11] | 16 [13 to 20]
Statistical Analysis 1: Comparison: Acyline Plus Placebo vs Acyline Plus 15 IU hCG vs Acyline Plus 60 IU hCG vs Acyline Plus 125 IU hCG; Test type: Superiority or Other; p < 0.05, ANOVA; Correlations between serum hormone levels and IT hormones, and between IT hormones were performed on 23 subjects in 4 groups using Spearmen technique

2. Primary Outcome: Serum Luteinizing Hormone (LH)
Time Frame: 10 days
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Acyline Plus Placebo | Acyline Plus 15 IU hCG | Acyline Plus 60 IU hCG | Acyline Plus 125 IU hCG | Acyline Plus Testosterone Gel
Number analyzed (Participants) | 6 | 7 | 5 | 5 | 8
IU/L | 0.13 [0.07 to 0.23] | 0.28 [0.2 to 1.63] | 0.49 [0.16 to 1.3] | 0.39 [0.28 to 1.7] | 0.14 [0.05 to 0.62]

3. Primary Outcome: Serum Follicle Stimulating Hormone (FSH)
Time Frame: 10 days
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Acyline Plus Placebo | Acyline Plus 15 IU hCG | Acyline Plus 60 IU hCG | Acyline Plus 125 IU hCG | Acyline Plus Testosterone Gel
Number analyzed (Participants) | 6 | 7 | 5 | 5 | 8
IU/L | 0.41 [0.17 to 0.46] | 0.41 [0.27 to 0.6] | 0.29 [0.24 to 1.0] | 0.28 [0.25 to 1.1] | 0.21 [0.18 to 0.27]

4. Primary Outcome: Intratesticular Testosterone (ITT-T)
Time Frame: 10 days
Measure: Median (Inter-Quartile Range); unit: IU/L
Arm/Group | Acyline Plus Placebo | Acyline Plus 15 IU hCG | Acyline Plus 60 IU hCG | Acyline Plus 125 IU hCG | Acyline Plus Testosterone Gel
Number analyzed (Participants) | 6 | 7 | 5 | 5 | 8
IU/L | 77 [40 to 223] | 136 [79 to 258] | 319 [139 to 2455] | 987 [895 to 1250] | 73 [34 to 264]

ADVERSE EVENTS:
Time Frame: overall study (1 year, 5 months)
Description: The first subject was screened 3/17/09; the last subject exited 8/17/10. Subjects in the study are asked about adverse events and concomitant medications at every visit.
Arm/Group | Acyline Plus Placebo | Acyline Plus 15 IU hCG | Acyline Plus 60 IU hCG | Acyline Plus 125 IU hCG | Acyline Plus Testosterone Gel
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7 | 0/5 | 0/5 | 0/8
Other Adverse Events (participants affected / at risk) | 1/6 | 1/7 | 3/5 | 2/5 | 1/8
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyline Plus Placebo (N=6) | Acyline Plus 15 IU hCG (N=7) | Acyline Plus 60 IU hCG (N=5) | Acyline Plus 125 IU hCG (N=5) | Acyline Plus Testosterone Gel (N=8)
hot flashes (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
dry itchy skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — dry itchy skin at site of gel application
fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — fatigue for 12 days
decreased libido (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
testicular soreness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
slight dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes